CLINICAL TRIAL: NCT05209698
Title: Health Outcomes in Patients With Parkinson's Disease in Israel: Associations With Accessibility, Utilization of Healthcare Services and Patients' Attitudes Among Different Ethnic Groups.
Brief Title: Self-Management Behaviors of Arabs and Jews With Parkinson's Disease and Their Associations With Health Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: 0128-19-COM1
Record Dates: First submitted 2022-01-23; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Parkinson Disease; Neuro-Degenerative Disease; Movement Disorders
Keywords: Self-management; Patient activation; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ethnic groups- Jews and Arabs: Data will be extracted from electronic medical records for all people with PD residing in a specific HMO district according to a record-based survey (e.g., individuals whose medical records include a diagnosis of PD). Currently, there are 2500 patients with PD in that district. In the second part of the study, a sub-sample of 100 Jewish and 100 Arab Patients with Parkinson's disease will be asked to answer standardized questionnaires.

SUMMARY:
The study will examine the reciprocal relationships between the community, healthcare system, and personal determinants of self-management behaviors in persons with Parkinson's disease and their association with the performance of these behaviors in persons with Parkinson's Disease.

In the first part of the study, data will be extracted from electronic medical records of 2500. In the second part of the study, a sub-sample of 200 participants with Parkinson's disease will be asked to answer standardized questionnaires.

DETAILED DESCRIPTION:
Parkinson's disease is a chronic, protracted condition. Its diverse symptoms affect the daily functioning and quality of life of patients and their families. The progressive disability is accompanied by medical complications and hospitalizations, which increase the economic burden on patients and healthcare systems. Factors that can mitigate these adverse consequences include care from a neurologist, rehabilitative treatments, and patients' use of self-management strategies. However, studies suggest that Patients with Parkinson from minority groups are less likely to be treated by a neurologist. Also, it is unclear whether Patients with Parkinson from minority groups are offered self-management strategies.

The study objectives were: To (1) to identify the reciprocal relationships among extra- and intra-personal level determinants of Self-Management Behaviors and their association with performance of these behaviors in persons with Parkinson's Disease, (2) identify the relationships between self-management behaviors (medical and lifestyle), function, and quality of life in patients with Parkinson's Disease.

Phase A of the study is a retrospective study based on extraction and analysis of data from electronic medical records, and phase B of the study is a cross-sectional study based on face-to-face meetings with a subsample of the patients whose data are included in the retrospective study.

ELIGIBILITY:
Inclusion Criteria for the retrospective study: People diagnosed with Parkinson's Disease.

Exclusion Criteria: None.

Inclusion Criteria for the cross-sectional study:

1. Diagnosis of PD.
2. Jewish sector will be fluency in Hebrew (comprehension, speaking, and reading), and for the Arab sector, fluency in Arabic or Hebrew (comprehension, speaking, and reading).

Exclusion Criteria for the cross-sectional study:

1. Acute hospitalization in the last 3 months.
2. Severe co-morbidities other than PD that affect daily living, special populations including pregnant women, minors (<18 years old).
3. Patients who are not eligible to sign consent forms due to physical or mental conditions.
4. People who have a guardian, score less than 20 in the Mini-Mental state exam test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PD within a distinct district of an HMO company have Parkinson's disease.
  Currently, there are 2,500 Patients with Parkinson's Disease in that district, of whom 281 are members of the Arab society.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Visits to a neurologist | 1 year
  extraction and analysis of data from Clalit's electronic medical records (EMR) of 2500 patients with Parkinson's Disease
Use of physical therapy services | 1 year
  extraction and analysis of data from Clalit's electronic medical records (EMR) of 2500 patients with Parkinson's Disease
Patient's Activation Measure (PAM-13®, Insignia Health) | 1 hour
  Patient activation' describes the skills, confidence and knowledge a person has in managing her/his own health and health care.
  It consists of 13 statements rated on a four-point Likert scale of level of agreement. The PAM-13 score is transformed into a 0-100 continuous scale according to a licensed conversion table (Insignia Health).
International Physical Activity Questionnaire- IPAQ-SHORT | 1 hour
  This questionnaire asks individuals to assess the number of days and amount of time they spent in the last 7 days in four categories: 1) vigorous activity (heavy lifting, aerobics, fast bicycling), 2) moderate activity (light lifting, moderate bicycling), 3) walking (at least 10 minutes), 4) sitting (watching TV, reading). Total physical activity is calculated as the sum of Walking + Moderate + Vigorous metabolic equivalent (MET) minutes/week scores.
Parkinson's Disease Questionnaire-39 (PDQ-39) | 1 hour
  This 39-item questionnaire is a patient-reported measure of health status and quality of life. It assesses how often people affected by PD experience difficulties across 8 dimensions of daily living, including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and wellbeing.
Nottingham Extended Activities of Daily Living (NEADL) | 1 hour
  The NEADL is a patient-reported outcome measure that consists of 22 items of everyday activities. It assesses patients' independence in activities of daily living.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Kafri, PhD, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Aba Hushi, Israel

REFERENCES:
- [Derived] Naamneh-Abuelhija B, Kafri M, Kestenbaum M, Giveon S, Kamah S, Shved S, Yogev-Seligmann G. Concealment of Parkinsons disease prevalence and impact on health and quality of life. Sci Rep. 2025 Mar 4;15(1):7551. doi: 10.1038/s41598-025-91579-8. PMID 40038366